CLINICAL TRIAL: NCT05295550
Title: Reliability of the Smartphone Inclinometer Application and Flexicurve on Thoracic Kyphosis
Brief Title: Reliability of the Smartphone Inclinometer App and Flexicurve
Acronym: Sİ-FC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gaziantep Islam Science and Technology University (Other)
Responsible Party: Principal Investigator, Gönül Elpeze, Master of Physiotherapy Physicaltherapist, Hasan Kalyoncu University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: HKU-GE-SPFC-Realiability
Record Dates: First submitted 2022-03-03; First posted 2022-03-25 (Actual); Last update posted 2025-09-02 (Actual); Status verified 2025-08

CONDITIONS: Disorder; Kyphosis Deformity of Thoracic Spine
MeSH Terms: conditions — Disease

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Flexicurve-Smartphone İnclinometer Application (Experimental): Measurement of thoracic kyphosis
  Interventions: Other: Realibility

INTERVENTIONS:
Other: Realibility — measurement of the thoracic kyphosis with flexicurve and Smartphone inclinometer app
  Other Names: İntra rater and inter rater

SUMMARY:
The presedent study evaluates intra-rater and inter-rater reliability of the Smartphone inclinometer app and the flexicurve, on the thoracic kyphosis

DETAILED DESCRIPTION:
Sixty subjects ranging from 17to 24 years of age were evaluated by two independent evaluators using the Flexicurve and the Smartphone inclinometer app to measure thoracic kyphosis

ELIGIBILITY:
Inclusion Criteria:

* over 30 degree toracic kyphosis,
* 18-30 age year old,
* individuals to willing participate in the study

Exclusion Criteria:

* Skolyoz (Cobb angle 10< ),
* rigid thoracic kyphosis,
* congenital spine disease,
* training with professional sports

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
İntra-İnterrater reliability fleksicurve and smartphone inclinometer app on thoracic kyphosis | 1 Year
  60 participant (35 male, 25 female) who have over 30 degree thoracic kyphosis were evaluated by two raters for finding correlation between flexicurve and smartphone inclinometer app.

CONTACTS AND LOCATIONS:
Overall Officials: GÖNÜL ELPEZE, Principal Investigator — HKU
Locations (1):
- Hasan Kalyoncu Üniversitesi, Şehitkamil, Gazi̇antep, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No